CLINICAL TRIAL: NCT06164665
Title: Effects of Pioglitazone on Exogenous Carbohydrate Oxidation During Steady-State Exercise at High Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22-07H
Record Dates: First submitted 2023-09-19; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: High Altitude
MeSH Terms: conditions — Altitude Sickness | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: randomized crossover placebo controlled double blinded study
Who Masked: Participant, Investigator
Masking Description: Treatment type (PIO/PLA) will be coded to de-identify treatment (Example: treatment A and treatment B or similar) to blinded staff. Assigned unblinded staff, responsible for administering the treatment to volunteers, will be responsible for creating treatment codes to match treatment. They will maintain record of randomization scheme and treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pioglitazone (Active Comparator): Pioglitazone administered as a 15 mg oral dose per day for 5 days
  Interventions: Drug: Pioglitazone 15mg
- Placebo (Placebo Comparator): Microcrystalline cellulose pill administered as an oral dose per day for 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pioglitazone 15mg — Pioglitazone (PIO) will be administered as a 15 mg oral dose per day for 5 days
  Other Names: Actos
  Arms: Pioglitazone
Other: Placebo — 100% microcrystalline cellulos
  Arms: Placebo

SUMMARY:
Apparent hypoxia-induced insulin insensitivity along with alterations in glucose kinetics suggests reduction in glucose uptake by the peripheral tissue is a primary factor contributing to reductions in exogenous glucose oxidation at HA. As such, the primary objective of this study is to determine the ability of an insulin sensitizer (Pioglitazone, PIO) to enhance exogenous glucose oxidation and metabolic clearance rate during metabolically-matched, steady-state exercise during acute HA exposure compared to placebo (PLA) in native lowlanders. Secondary objective of this study will be to assess the impact of PIO on markers of inflammation and iron status compared to PLA. This randomized crossover placebo control double blinded study will examine substrate oxidation and glucose kinetic responses to ingesting supplemental carbohydrate (glucose) during metabolically-matched, steady-state exercise with acute (~5 h) exposure to HA (460 mmHg, or 4300m, barometric pressure similar to Pike's Peak) after receiving PIO (HA+PIO), or after receiving a matched placebo (HA+PLA). Eight healthy, recreationally active males between the ages of 18-39 yrs will be required to complete this study. Following a 4 day glycogen normalization period receiving PIO or PLA daily, volunteers will complete two 80-min trials, performing metabolically-matched, steady-state aerobic (same absolute workload corresponding to ~55 ± 5% of V̇O2peak at HA) exercise on a treadmill, and consuming 145 g of glucose (1.8 g/min); one trial with HA+PIO and the other with HA+PLA. A dual glucose tracer (13C-glucose oral ingestion and [6,6-2H2]-glucose primed, continuous infusion) technique and indirect calorimetry will be used to selectively analyze endogenous and exogenous glucose oxidation, as well as glucose rate of appearance (Ra), disappearance (Rd) and metabolic clearance rate (MCR). Serial blood samples will be collected during each trial to assess endocrine and circulating substrate responses to exercise, carbohydrate, and hypoxia with or without PIO. All trials will occur at the same time of day in the USARIEM hypobaric/hypoxic chamber and be separated by a minimum 10-d washout period. The primary risks associated with this study include those associated with acute hypobaric hypoxia, exercise, and blood sampling.

DETAILED DESCRIPTION:
This randomized crossover placebo controlled double blinded study will examine substrate oxidation and glucose kinetic responses to ingesting supplemental carbohydrate (glucose) during metabolically-matched, steady-state exercise with acute (~5 h) exposure to HA (460 mmHg) after short-term (5 days) use of Pioglitazone (HA+PIO), or matched placebo (HA+PLA). Eight healthy, recreationally active males between the ages of 18-39 yrs will be enrolled. Following a 48-hr muscle glycogen normalization period, volunteers will complete 80-min of metabolically-matched, steady-state (same absolute workload corresponding to ~55 ± 5% of V̇O2peak at HA) exercise on a treadmill, and consume 145 g of glucose (1.8 g/min) with HA+PIO and HA+PLA. A dual glucose tracer (13C-glucose oral ingestion and [6,6-2H2]-glucose primed, continuous infusion) technique and indirect calorimetry will be used to analyze endogenous and exogenous glucose oxidation, as well as glucose rate of appearance (Ra), disappearance (Rd), and MCR. Serial blood samples will be collected during each trial to assess endocrine and circulating substrate responses to exercise, carbohydrate, and hypoxia, with or without PIO. Isotope methodology and aerobic exercise protocols will be identical to our previous work (3, 4), allowing comparison of outcomes across studies. All trials will be conducted in the USARIEM hypobaric/hypoxic chamber and be separated by a minimum 10-d washout period.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 - 39 years
* Born at altitudes less than 2,100 m
* Physically active (exercise minimum 2 days per week)
* Have supervisor approval (permanent party military and civilians)
* Willing to refrain from alcohol, smokeless nicotine products and dietary supplement use during study periods
* Fully vaccinated against COVID-19

Exclusion Criteria:

* Born at altitudes greater than 2,100 m
* Musculoskeletal injuries that compromise exercise capability
* Metabolic or cardiovascular abnormalities, or gastrointestinal disorders
* Taking medication that affects macronutrient metabolism and/or the ability to participate in strenuous exercise
* Living in areas that are more than 1,200 m, or traveled to areas that are more than 1,200 m for five days or more within 2 months of data collection
* Evidence of apnea or other sleeping disorders
* Prior diagnosis of high altitude pulmonary edema or high altitude cerebral edema
* Presence of asthma or respiratory tract infections
* Smoking or vaping
* Taking medications that interfere with oxygen delivery and transport
* Anemia (HCT <38% and HBG <12.5 g/dL) and Sickle Cell Anemia/Trait
* Blood donation within 8 weeks of beginning the study
* Unwilling or unable to consume study diets or foods provided due to personal preference, dietary restrictions, and/or food allergies
* Unwilling or unable to adhere to study physical restrictions

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of Exogenous Glucose Oxidation | 8 hours
  Determine the effects of PIO on exogenous glucose oxidation and glucose turnover during exercise under acute HA exposure compared to PLA

SECONDARY OUTCOMES:
Concentration of Interleukin-6 | 8 hours
  Determine the effects of PIO on inflammation during acute HA exposure compared to PLA.
Concentration of Serum Iron | 8 hours
  Determine the effects of PIO on markers of iron status during acute HA exposure compared to PLA

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT06164665/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT06164665/ICF_001.pdf